CLINICAL TRIAL: NCT07289087
Title: A Real-World Observational Study on Patient-Reported Outcomes in Allogeneic Stem Cell Transplantation (Allo-SCT) and CAR-T Therapy
Brief Title: Patient-Reported Outcomes in Allogeneic Stem Cell Transplantation and CAR-T Therapy
Acronym: QOL-ONE PRO-CT
Status: Not yet recruiting | Type: Observational
Sponsor: Associazione Qol-one (Other)
Responsible Party: Sponsor
Other Study IDs: QOL-ONE PRO-CT
Record Dates: First submitted 2025-11-17; First posted 2025-12-17 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Quality of Life; Patient Reported Outcome (PRO); Allogeneic Blood and Marrow Transplantation (BMT); CAR T Cell Therapy
Keywords: Quality of Life; CAR-T cell therapy; Allogenic BMT; Patient Reported Outcome; Leukemia; Multiple Myeloma; Lymphoma
MeSH Terms: conditions — Leukemia; Multiple Myeloma; Lymphoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- CAR-T
- ALLO-SCT

SUMMARY:
3.1. Overview Prospective, multicenter, observational cohort study comparing short-term PROs measured with the HM-PRO between two exposure groups: patients undergoing allogeneic stem cell transplantation (allo-SCT) and patients receiving CAR-T cell therapy. Patients will be enrolled at hospital admission for the index inpatient procedure and followed through the inpatient stay (admission → discharge). The study is non-randomized and designed to describe trajectories of symptoms and HRQoL and to estimate the between-group difference in deterioration of HM-PRO scores (primary estimand: mean difference in change score, CAR-T vs allo-SCT).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with a hematologic malignancy (e.g., leukemia, lymphoma, multiple myeloma)
* Undergoing either allogeneic SCT or CAR-T therapy
* Able and willing to provide written informed consent
* Sufficient Italian proficiency to complete the HM-PRO
* Signed informed consent

Exclusion Criteria:

* Cognitive or physical impairments that preclude the ability to complete questionnaires
* Estimated life expectancy < 7 days at the time of admission

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults (≥18 years) with a hematologic malignancy admitted for either (a) allo-SCT or (b) CAR-T cell therapy.
Sampling Method: Probability Sample
Enrollment: 162 (Estimated)
Dates: Start 2026-02-15 (Estimated); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
To assess and compare short-term patient-reported outcomes [PROs (symptom burden and QoL impact)] between patients receiving allo-SCT and CAR-T therapy using the HM-PRO questionnaire (Impact Scale, Symptoms Scale) from admission to hospital discharge | 3 MONTHS
  The primary outcome aims to evaluate the impact of CAR-T therapy and allogeneic transplantation on patients' quality of life using a specific questionnaire (HM-PRO), which assesses PROs (quality of life and symptoms) in hematologic patients, with the goal of determining whether there are differences between the two patient groups.
  In the HM-PRO questionnaire values range from 0 to 100. Lower values correspond to a better quality of life and a lower symptom burden.

SECONDARY OUTCOMES:
To describe PRO trajectories during hospitalization | 3 MONTHS
  Patient-reported outcomes will be assessed using the Hematological Malignancy Patient-Reported Outcome (HM-PRO) instrument, which includes an Impact Scale and a Symptoms Scale. HM-PRO assessments will be performed at five predefined time points during hospitalization: T1 (hospital admission), T2 (day of infusion), T3 (day 3 post-infusion), T4 (day 10 post-infusion), and T5 (day of discharge). The secondary outcome will describe within-patient trajectories of HM-PRO scores over these time points. Data will be summarized using mean scores and mean changes from baseline (T1) for total and domain scores, to characterize changes in symptom burden and QoL impact throughout hospitalization.
To assess differences in PROs based on disease type (e.g., Leukemia, lymphoma, myeloma) | 3 MONTHS
  Since patients with different hematologic diseases are involved, the quality-of-life and symptom outcomes may vary for each condition.
To assess differences in PROs based on disease status (remission vs progression) | 3 MONTHS
  Patients at enrollment may be in remission or in disease progression. the quality-of-life and symptom outcomes may vary for each condition.
To assess differences in PROs based on treatment line (first-line vs multiple lines) | 3 MONTHS
  At enrollment, patients may have received first vs multiple lines of treatment. the quality-of-life and symptom outcomes may vary for each condition.
To validate the use of the HM-PRO in the context of inpatient care for advanced therapies. | 3 MONTHS
  This outcome will evaluate the psychometric properties of the Hematological Malignancy Patient-Reported Outcome (HM-PRO) questionnaire in the inpatient setting of advanced cellular therapies (allo-SCT and CAR-T). HM-PRO assessments are collected at five time points during hospitalization-T1 (admission), T2 (day of infusion), T3 (day 3 post-infusion), T4 (day 10 post-infusion), and T5 (discharge). Psychometric analyses will assess:
  Internal consistency reliability of the Impact and Symptoms Scales (Cronbach's alpha).
  Construct validity, evaluated through known-groups comparisons (allo-SCT vs CAR-T; remission vs progression).
  Responsiveness to clinical change, assessed by changes in HM-PRO scores over time in relation to clinical status and adverse events.
  These analyses will determine whether HM-PRO performs adequately for use in routine inpatient clinical practice for advanced therapies.

DOCUMENTS (1):
  • Study Protocol (2025-10-06): https://cdn.clinicaltrials.gov/large-docs/87/NCT07289087/Prot_000.pdf